CLINICAL TRIAL: NCT05059457
Title: A Pilot to Asses Hemoglobin Concentration Obtained From Capillary and Venous Blood Measured Using the HemoCue 201+ Hemoglobin Analyzer in a Controlled and Field Setting
Brief Title: Comparison of Blood Sampling Methods for Hemoglobin Measurement
Status: Completed | Type: Observational
Sponsor: ICF Macro, Inc. (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Uganda Bureau of Statistics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 720-OAA-18C-00083
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Anemia
Keywords: Anemia; DHS surveys; Point-of-care; Hemoglobin; Survey methods
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Controlled setting: single capillary and pooled capillary and venous blood: Single drop capillary blood, pooled capillary blood, and venous blood will be collected and hemoglobin measured among non-pregnant women age 15-49 and children age 6-59 months in a controlled setting.
  Interventions: Device: Blood source: single and pooled capillary and venous blood
- Field setting: single capillary and venous blood: Single drop capillary blood and venous blood will be collected and hemoglobin measured among non-pregnant women age 15-49 and children age 6-59 months in a field setting.
  Interventions: Device: Blood source: single capillary and venous blood
- Field setting: pooled capillary and venous blood: Pooled capillary blood and venous blood will be collected and hemoglobin measured among non-pregnant women age 15-49 and children age 6-59 months in a field setting.
  Interventions: Device: Blood source: pooled capillary and venous blood

INTERVENTIONS:
Device: Blood source: single and pooled capillary and venous blood — * A single drop of capillary blood (blood drop #3) will be placed in a microcuvette directly from a finger/heel and tested using a HemoCue 201+.
  * Pooled capillary blood will be placed in a Microtainer® tube (250-500 µL) containing EDTA and then a drop of blood placed in a microcuvette and tested using a HemoCue 201+.
  * Venous blood will be collected into a 3mL Vacutainer tube containing EDTA and then a drop of blood will be placed in a microcuvette and tested using a HemoCue 201+ and autoanalyzer.
  Groups: Controlled setting: single capillary and pooled capillary and venous blood
Device: Blood source: single capillary and venous blood — * A single drop of capillary blood (blood drop #3) will be placed in a microcuvette directly from a finger/heel and tested using a HemoCue 201+ .
  * Venous blood will be collected into a 3mL Vacutainer tube containing EDTA and then a drop of blood will be placed in a microcuvette and tested using a HemoCue 201+ and autoanalyzer.
  Groups: Field setting: single capillary and venous blood
Device: Blood source: pooled capillary and venous blood — * Pooled capillary blood will be placed in a Microtainer® tube (250-500 µL) containing EDTA and then a drop of blood placed in a microcuvette and tested using a HemoCue 201+.
  * Venous blood will be collected into a 3mL Vacutainer tube containing EDTA and then a drop of blood will be placed in a microcuvette and tested using a HemoCue 201+ and autoanalyzer.
  Groups: Field setting: pooled capillary and venous blood

SUMMARY:
This study is designed to inform The DHS Program on whether there are variations in hemoglobin concentration using the DHS standard technique of a single drop of capillary blood and alternative blood sources (pooled capillary and venous blood) using the HemoCue 201+ analyzer compared to venous blood using a clinical hematology autoanalyzer.

Research Objectives:

1. To determine if there are differences in the hemoglobin concentration between a single drop of capillary blood (blood drop #3) and a pooled drop of capillary blood measured on the HemoCue 201+ analyzer in apparently healthy non-pregnant women age 15-49 and children age 6-59 months in a controlled setting (i.e., blood specimens are collected in a laboratory setting).
2. To determine if there are differences in the hemoglobin concentration between a single drop of capillary blood (blood drop #3) measured on the HemoCue 201+ analyzer against venous blood measured on HemoCue 201+ analyzer and a clinical autoanalyzer in apparently healthy non-pregnant women age 15-49 and children age 6-59 months in a controlled and field setting.
3. To determine if there are differences in the hemoglobin concentration between a pooled drop of capillary blood measured on the HemoCue 201+ analyzer against venous blood measured on HemoCue 201+ analyzer and a clinical autoanalyzer in apparently healthy non-pregnant women age 15-49 and children age 6-59 months in a controlled and field setting.
4. To compare results of hemoglobin distribution and estimates of anemia prevalence using two types of capillary blood (single drop and pooled) and venous blood measured on the HemoCue 201+ analyzer and a clinical autoanalyzer using venous blood in a controlled and field setting.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-59 months or non-pregnant women 15-49
* Apparently healthy individuals
* Consent to participate in the study

Exclusion Criteria:

* Children less than 6 months or over 59 months
* Women less than 15 years of age or greater than 49 years of age
* Pregnant women

Ages: 6 Months to 49 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants will be children 6-59 months and non-pregnant women 15-49 years. In the controlled setting, participants will be selected from nearby communities and brought to the Ebenezer Lab in Kampala, Uganda. In the field setting, participants will be selected from households eligible for the DHS-8 questionnaire pilot in districts located near Kampala, Uganda.
Sampling Method: Probability Sample
Enrollment: 1082 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-09-26 (Actual)

PRIMARY OUTCOMES:
Hemoglobin measurement | Day 1
  Difference (correlation, concordance, paired t-test) in hemoglobin concentration between each blood source measured with the HemoCue 201+ compared to venous blood measured with a clinical autoanalyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Sorrel ML Namaste, DrPH, Principal Investigator — ICF
Locations (2):
- Uganda (2):
  - Ebenezer Lab, Kampala
  - Uganda Bureau of Statistics, Kampala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Namaste SM, Baingana R, Brindle E. Hemoglobin measurement in venous blood compared with pooled and single-drop capillary blood: a method-comparison study in a controlled and survey setting in Uganda among children and women. Am J Clin Nutr. 2024 Apr;119(4):949-959. doi: 10.1016/j.ajcnut.2023.12.025. Epub 2024 Jan 3. PMID 38176682